CLINICAL TRIAL: NCT05552508
Title: BURAN: Effects of Benralizumab on Airway Dynamics in Severe Eosinophilic Asthma Using Functional Respiratory Imaging Parameters
Brief Title: BURAN: Benralizumab on Airway Dynamics in Severe Eosinophilic Asthma Using Functional Respiratory Imaging
Acronym: BURAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3250R00107; 2022-000152-11 (EudraCT Number)
Record Dates: First submitted 2022-04-27; First posted 2022-09-23 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Asthma
Keywords: BURAN; Inhaled Corticosteroids; Long-acting β2 agonists; Benralizumab; Eosinophilic Asthma
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — benralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Benralizumab (Experimental): Participants will receive 3 doses of benralizumab having a strength of 30 mg subcutaneously once every 4 weeks (Week 0, Week 4, and Week 8).
  Interventions: Combination Product: Benralizumab

INTERVENTIONS:
Combination Product: Benralizumab — Participants will receive benralizumab subcutaneously.
  Other Names: Fasenra

SUMMARY:
This study will assess the effects of benralizumab on airway dynamics in severe eosinophilic asthma in terms of quantitative computed tomography (CT)-derived measurements of pulmonary structure and function using the Functional Respiratory Imaging (FRI) platform.

DETAILED DESCRIPTION:
This is a phase IV, interventional single group, open-label, uncontrolled, prospective, multicenter clinical trial.

This study will be conducted in male and female participants ≥18 years old with established severe eosinophilic asthma as defined by European Respiratory Society (ERS)/American Thoracic Society (ATS) clinical guidelines inadequately controlled by treatment with Inhaled Corticosteroids-Long-acting β2 agonists (ICS-LABA) with or without oral corticosteroids (OCS) or other asthma controller medications.

Each participant will participate in the study for a minimum of 15 weeks and up to 23 weeks.

This study will comprise of:

Screening visit (V0) Visit 1 (V1; week 0; within 1 to 21 days of screening) Visit 2 (V2; week 4 ± 5 days) Visit 3 (V3; week 8 ± 5 days) Visit 4 (V4; week 13 ± 5 days) Follow-up (2 weeks [± 7 days] after V4) - Phone call follow-up. Participants will be discharged from the study after the phone call follow-up is completed.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are diagnosed with asthma with documented reversibility post-bronchodilator or salbutamol either historical or at Visit 0 (V0).
* Participants who have documented treatment with ICS and LABA for ≥ 3 months prior to V0 with or without oral corticosteroids and additional asthma controllers.
* Participants who have documented peripheral blood eosinophil count ≥ 300 cells/μL at V0, or if Oral Corticosteroids (OCS)-dependent, a documented peripheral blood eosinophil count ≥ 150 cells/μL at V0.
* Participants who have had a minimum of 2 exacerbations in the last 12 months prior to V0.
* Participants who have pre-bronchodilator Forced Expiratory Volume in 1 second (FEV1)/Forced Vital Capacity (FVC) ≤ 70% at Visit 0 (V0).
* Participants who have pre-bronchodilator Forced Expiratory Volume in 1 second (FEV1) < 80% of predicted at V0.
* Participants who can perform acceptable and repeatable spirometry.
* Participants who can withhold asthma maintenance medication for at least 12 hours prior to V0, 1 and 4 where spirometry and/or Computed Tomography (CT) scan procedures will be performed except for once-a-day dosage where 24 hours will be required.
* Female participants who have a negative pregnancy test prior to administration of the investigational product (IP) and high-resolution CT scan and must agree to use a highly effective method of birth control from randomization throughout the study duration and within 12 weeks after last dose of IP.

Exclusion Criteria:

* Participants who are unstable or who experienced an exacerbation/infection in the 6 weeks before V0.
* Participants with acute upper or lower airway infection in the 6 weeks before V0.
* Participants diagnosed with clinically important pulmonary disease other than asthma, or participants who have ever been diagnosed with pulmonary or systemic disease, other than asthma that are associated with elevated peripheral eosinophil count.
* Receipt of any biologic products for asthma within 4 months or 5 half-lives prior to V0 whichever is longer.
* History or current use of chronic (i.e., > 4 weeks) immunosuppressive medication.
* History of lung volume reduction surgery, lung resection, thermal bronchoplasty at any time before visit 0 (V0) or on active phase of pulmonary rehabilitation.
* Participants with current malignancy or history of malignancy.
* History of other clinically significant disease or abnormality.
* Participants with positive Hepatitis B, C or HIV.
* Participants with:

Positive COVID-19 test at V0, COVID-19 disease within 6 weeks before V0 or History of severe COVID-19 disease at any time, defined by the need for Intensive Care Unit stay or Mechanical Ventilation (invasive or non-invasive).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (10):
  - Research Site, Walnut Creek, California
  - Research Site, Loxahatchee Groves, Florida
  - Research Site, Plantation, Florida
  - Research Site, Greenwood, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, St Louis, Missouri
  - Research Site, DuBois, Pennsylvania
  - Research Site, Tyler, Texas
  - Research Site, Webster, Texas
  - Research Site, Charlottesville, Virginia
- Australia (2):
  - Research Site, Clayton
  - Research Site, Toorak Gardens
- Belgium (2):
  - Research Site, Liège
  - Research Site, Namur
- Research Site, Montpellier, France
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Santander
  - Research Site, Villarreal (Castellón)
- United Kingdom (2):
  - Research Site, Bradford
  - Research Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Genofre E, Carstens D, DeBacker W, Muchmore P, Panettieri RA Jr, Rhodes K, Shih VH, Trudo F. The effects of benralizumab on airway geometry and dynamics in severe eosinophilic asthma: a single-arm study design exploring a functional respiratory imaging approach. Respir Res. 2023 May 3;24(1):121. doi: 10.1186/s12931-023-02415-4. PMID 37131265
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00107&attachmentIdentifier=1a0d1d2c-2695-4f84-9590-a6ea603f3755&fileName=D3250r00107_(264960)-CSP-Final-_Redacted_1.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00107&attachmentIdentifier=f4729df0-fdab-4ed7-b0b6-15902639c375&fileName=D3250r00107_(264960)-CSR_Synopsis_Final-Redacted_1.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00107&attachmentIdentifier=3363bf1b-9b8b-4293-b6b6-b7b78a29cd0f&fileName=D3250r00107_(264960)-SAP_Final-Redacted_1.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 11 October 2022 to 19 July 2024 at 24 study centers in in Australia, Belgium, France, Portugal, Spain, United Kingdom, and United States.
Pre-assignment Details: Participants who met the inclusion criteria and none of the exclusion criteria were enrolled to the study. Informed Consent Form (ICF) was signed prior of screening procedures. All study assessments were performed as per the Schedule of Activities.
Groups:
- Benralizumab: Participants received 3 doses of benralizumab 30 milligrams (mg) as subcutaneous injection once every 4 weeks (Week 0, Week 4, and Week 8).
Period: Overall Study
Arm/Group | Benralizumab
Started | 45
Completed | 42
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: Primary analysis population set consisted portion of the evaluable population that did not have any acute asthma exacerbation nor lower respiratory tract infection during the study period.
Groups:
- Benralizumab: Participants received 3 doses of benralizumab 30 mg as subcutaneous injection once every 4 weeks (Week 0, Week 4, and Week 8).
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Untrimmed Total Mucus Volume at TLC
Description: Change from baseline in airway dynamics after 13 weeks following treatment with benralizumab, using total mucus volume (specific airway volume) at total lung capacity (TLC) measurements from untrimmed airways was assessed.
Time Frame: Baseline and Week 13
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
Milliliters (mL)
  All participants | -0.1279 (0.4199)
  Participants with >=4 mucus plugs: number analyzed (Participants) | 27
  Participants with >=4 mucus plugs | -0.1822 (0.4977)
  Participants with <4 mucus plugs: number analyzed (Participants) | 12
  Participants with <4 mucus plugs | -0.0056 (0.0111)
  OCS-dependent participants: number analyzed (Participants) | 2
  OCS-dependent participants | -0.1619 (0.4627)
  Non-OCS-dependent participants: number analyzed (Participants) | 37
  Non-OCS-dependent participants | -0.1260 (0.4244)
Statistical Analysis 1: Comparison: Benralizumab; All participants; Test type: Other; p = 0.0327, t-test, 2 sided
Statistical Analysis 2: Comparison: Benralizumab; Participants with >=4 mucus plugs; Test type: Other; p = 0.0359, t-test, 2 sided
Statistical Analysis 3: Comparison: Benralizumab; Participants with <4 mucus plugs; Test type: Other; p = 0.1088, t-test, 2 sided
Statistical Analysis 4: Comparison: Benralizumab; Non-OCS-dependent participants; Test type: Other; p = 0.0391, t-test, 2 sided

2. Secondary Outcome: Change From Baseline in Untrimmed Total Mucus Plugs Score at TLC
Description: Change from baseline in untrimmed total mucus plugs score at TLC was assessed. Mucus plugs was scored with a scoring system similar to that by Dunican et al. with the Severe Asthma Research Program (SARP) based on bronchopulmonary segmental anatomy. The mucus score was calculated by counting the number of bronchopulmonary segments which contained 1 or more mucus plug, up to a maximum score of 18 corresponding to the 18 bronchopulmonary segments present in most people. In this system, a mucus plug is defined as a complete occlusion of the airway visible at TLC. Each bronchopulmonary segment is given a score of 1 (mucus plug[s] present) or 0 (mucus plug[s] absent). The segment scores of each lobe are summed to generate a total mucus score for both lungs, yielding a mucus score ranging from 0-18. Higher scores indicate worse outcome.
Time Frame: Baseline and Week 13
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
Scores on a scale | -11.0 (32.8)
Statistical Analysis 1: Comparison: Benralizumab; Test type: Other; p = 0.0423, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Untrimmed Total Air Trapping at FRC
Description: Change from baseline in untrimmed total air trapping at FRC was assessed.
Time Frame: Baseline and Week 13
Population: Primary analysis population set consisted portion of the evaluable population that did not have any acute asthma exacerbation nor lower respiratory tract infection during the study period. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of air trapping
Arm/Group | Benralizumab
Number analyzed (Participants) | 34
Percentage of air trapping | -0.1410 (12.1660)
Statistical Analysis 1: Comparison: Benralizumab; Test type: Other; p = 0.9465, t-test, 2 sided

4. Secondary Outcome: Change From Baseline in Trimmed Distal Airway Wall Volume at TLC
Description: Change from baseline in trimmed distal airway wall volume at TLC was assessed. Change from baseline in airway dynamics at Week 13 following treatment with benralizumab as measured by secondary FRI endpoints, irrespective of participants characteristics was assessed.
Time Frame: Baseline and Week 13
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
mL | -0.9386 (6.1359)
Statistical Analysis 1: Comparison: Benralizumab; Test type: Other; p = 0.3455, t-test, 2 sided

5. Secondary Outcome: Change From Baseline in Untrimmed Distal Airway Volume at TLC
Description: Change from baseline in untrimmed distal airway volume at TLC was assessed.
Time Frame: Baseline and Week 13
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
mL | 1.1225 (4.5836)
Statistical Analysis 1: Comparison: Benralizumab; Test type: Other; p = 0.2484, t-test, 2 sided

6. Secondary Outcome: Change From Baseline in Untrimmed Distal Airway Volume at Functional Residual Capacity (FRC)
Description: Change from baseline in untrimmed distal airway volume at FRC was assessed.
Time Frame: Baseline and Week 13
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Benralizumab
Number analyzed (Participants) | 34
mL | 0.5079 (1.9741)
Statistical Analysis 1: Comparison: Benralizumab; Test type: Other; p = 0.9405, t-test, 2 sided

7. Secondary Outcome: Change From Baseline in Untrimmed Total Lung Volume at TLC
Description: Change from baseline in untrimmed total lung volume at TLC was assessed.
Time Frame: Baseline and Week 13
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
Liters (L) | 0.0287 (0.4416)
Statistical Analysis 1: Comparison: Benralizumab; Test type: Other; p = 0.6867, t-test, 2 sided

8. Secondary Outcome: Change From Baseline in Untrimmed Total Lung Volume at FRC
Description: Change from baseline in untrimmed total lung volume at FRC was assessed.
Time Frame: Baseline and Week 13
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Benralizumab
Number analyzed (Participants) | 34
Liters (L) | -0.0275 (0.5101)
Statistical Analysis 1: Comparison: Benralizumab; Test type: Other; p = 0.7554, t-test, 2 sided

9. Secondary Outcome: Correlation Between Untrimmed Total Mucus Volume Measured at TLC and Pre-bronchodilator Forced Expiratory Volume in 1 Second (Pre-BD FEV1)
Description: The relationship between airway dynamics and conventional lung function measurements, cross sectionally (at week 0) and irrespective of participants characteristics was assessed. Positive correlations were identified by values greater than 0, and negative correlations were identified by values less than 0. Statistical significance is indicated when the lower limit of the 95% confidence interval (CI) for the correlation is greater than 0 for positive correlations or less than 0 for negative correlations.
  Here, "Number" in measure type is indicating data of Spearman's rank correlation coefficient.
Time Frame: At Baseline (Week 0)
Population: Baseline endpoints analysis set included all participants who had baseline measurements and who had at least one dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 43
Correlation coefficient | -0.2710 [-0.5260 to 0.0352]

10. Secondary Outcome: Correlation Between Untrimmed Total Mucus Plugs Score at TLC and Pre-BD FEV1
Description: The relationship between airway dynamics and conventional lung function measurements, cross sectionally (at week 0) and irrespective of participants characteristics was assessed. Positive correlations were identified by values greater than 0, and negative correlations were identified by values less than 0. Statistical significance is indicated when the lower limit of the 95% CI for the correlation is greater than 0 for positive correlations or less than 0 for negative correlations.
  Here, "Number" in measure type is indicating data of Spearman's rank correlation coefficient.
Time Frame: At Baseline (Week 0)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 43
Correlation coefficient | -0.2795 [-0.5326 to 0.0260]

11. Secondary Outcome: Correlation Between Untrimmed Total Air Trapping at FRC and Pre-BD FEV1
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: Baseline endpoints analysis set included all participants who had baseline measurements and who had at least one dose of study intervention. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 40
Correlation coefficient | -0.6892 [-0.8210 to -0.4742]

12. Secondary Outcome: Correlation Between Trimmed Distal Airway Wall Volume at TLC and Pre-BD FEV1
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 42
Correlation coefficient | 0.5380 [0.2738 to 0.7205]

13. Secondary Outcome: Correlation Between Untrimmed Distal Airway Volume at TLC and Pre-BD FEV1
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: Baseline endpoints analysis set included all participants who had baseline measurements and who had at least one dose of study intervention. Here, 'number analyzed in each row' signifies the participants with available data that were analyzed for specified category.
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 43
Correlation coefficient | 0.6556 [0.4360 to 0.7958]

14. Secondary Outcome: Correlation Between Untrimmed Distal Airway Volume at FRC and Pre-BD FEV1
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 43
Correlation coefficient | 0.4357 [0.1383 to 0.6548]

15. Secondary Outcome: Correlation Between Untrimmed Total Lung Volume at TLC and Pre-BD FEV1
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 43
Correlation coefficient | 0.2122 [-0.0966 to 0.4799]

16. Secondary Outcome: Correlation Between Untrimmed Total Lung Volume at FRC and Pre-BD FEV1
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 43
Correlation coefficient | -0.1655 [-0.4519 to 0.1560]

17. Secondary Outcome: Correlation Between Untrimmed Total Mucus Volume Measured at TLC and Pre-bronchodilator Forced Vital Capacity (Pre-BD FVC)
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 43
Correlation coefficient | -0.0471 [-0.3421 to 0.2574]

18. Secondary Outcome: Correlation Between Untrimmed Total Mucus Plugs Score at TLC and Pre-BD FVC
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 43
Correlation coefficient | -0.0273 [-0.3247 to 0.2756]

19. Secondary Outcome: Correlation Between Untrimmed Total Air Trapping at FRC and Pre-BD FVC
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 40
Correlation coefficient | -0.3432 [-0.5886 to -0.0311]

20. Secondary Outcome: Correlation Between Trimmed Distal Airway Wall Volume at TLC and Pre-BD FVC
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 42
Correlation coefficient | 0.5476 [0.2863 to 0.7269]

21. Secondary Outcome: Correlation Between Untrimmed Distal Airway Volume at TLC and Pre-BD FVC
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 43
Correlation coefficient | 0.6110 [0.3742 to 0.7670]

22. Secondary Outcome: Correlation Between Untrimmed Distal Airway Volume at FRC and Pre-BD FVC
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 40
Correlation coefficient | 0.4706 [0.1806 to 0.6789]

23. Secondary Outcome: Correlation Between Untrimmed Total Lung Volume at TLC and Pre-BD FVC
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 43
Correlation coefficient | 0.4947 [0.2227 to 0.6891]

24. Secondary Outcome: Correlation Between Untrimmed Total Lung Volume at FRC and Pre-BD FVC
Description: as for outcome 10
Time Frame: At Baseline (Week 0)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Benralizumab
Number analyzed (Participants) | 40
Correlation coefficient | 0.1451 [-0.1761 to 0.4354]

25. Secondary Outcome: Change From Baseline in Untrimmed Total Mucus Volume Measured at TLC With and Without Adjustment for Pre-BD FEV1
Description: The relationship between changes from baseline (week 0) in airway dynamics and conventional lung function measurements at Week 13, after accounting for baseline measurements of conventional lung function was assessed with and without adjustment for conventional lung function measures (pre-BD FEV1).
Time Frame: Baseline and Week 13
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
mL
  No adjustment for pre-BD FEV1 | 0.05 [0.00 to 0.11]
  Adjusted for pre-BD FEV1 | 0.06 [0.00 to 0.12]

26. Secondary Outcome: Change From Baseline in Untrimmed Total Mucus Plugs Score at TLC With and Without Adjustment for Pre-BD FEV1
Description: Relationship between changes from baseline (week 0) in airway dynamics and conventional lung function measurements at Week 13, after accounting for baseline measurements of conventional lung function was assessed with and without adjustment for conventional lung function measures (pre-BD FEV1). Mucus plugs was scored with a scoring system similar to that by Dunican et al. with SARP based on bronchopulmonary segmental anatomy. Mucus score was calculated by counting number of bronchopulmonary segments which contained 1 or more mucus plug, up to a maximum score of 18 corresponding to the 18 bronchopulmonary segments present in most people. In this system, a mucus plug is defined as a complete occlusion of airway visible at TLC. Each bronchopulmonary segment is given a score of 1 (mucus plug present) or 0 (mucus plug absent). The segment scores of each lobe are summed to generate a total mucus score for both lungs, yielding a mucus score ranging from 0-18. Higher scores = worse outcome.
Time Frame: Baseline and Week 13
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
Scores on a scale
  No adjustment for pre-BD FEV1 | 4.38 [-2.87 to 11.63]
  Adjusted for pre-BD FEV1 | 5.97 [-1.75 to 13.69]

27. Secondary Outcome: Change From Baseline in Untrimmed Total Air Trapping at FRC With and Without Adjustment for Pre-BD FEV1
Description: as for outcome 25
Time Frame: Baseline and Week 13
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percentage of air trapping
Arm/Group | Benralizumab
Number analyzed (Participants) | 34
Percentage of air trapping
  No adjustment for pre-BD FEV1 | 3.18 [-3.65 to 10.01]
  Adjusted for pre-BD FEV1 | 5.24 [-1.23 to 11.71]

28. Secondary Outcome: Change From Baseline in Trimmed Distal Airway Wall Volume at TLC With and Without Adjustment for Pre-BD FEV1
Description: as for outcome 25
Time Frame: Baseline and Week 13
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
mL
  No adjustment for pre-BD FEV1 | 5.29 [-1.39 to 11.97]
  Adjusted for pre-BD FEV1 | 5.61 [-1.27 to 12.48]

29. Secondary Outcome: Change From Baseline in Untrimmed Distal Airway Volume With and Without Adjustment for Pre-BD FEV1
Description: as for outcome 25
Time Frame: Baseline and Week 13
Population: Primary analysis population set consisted portion of the evaluable population that did not have any acute asthma exacerbation nor lower respiratory tract infection during the study period. Here, 'number analyzed in each row' signifies the participants with available data that were analyzed for specified category.
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
mL
  Untrimmed distal airway volume at TLC: No adjustment for pre-BD FEV1 | 2.20 [-1.09 to 5.49]
  Untrimmed distal airway volume at TLC: Adjusted for pre-BD FEV1 | 0.61 [-2.65 to 3.88]
  Untrimmed distal airway volume at FRC: No adjustment for pre-BD FEV1: number analyzed (Participants) | 34
  Untrimmed distal airway volume at FRC: No adjustment for pre-BD FEV1 | -1.28 [-2.82 to 0.27]
  Untrimmed distal airway volume at FRC: Adjusted for pre-BD FEV1: number analyzed (Participants) | 34
  Untrimmed distal airway volume at FRC: Adjusted for pre-BD FEV1 | -1.52 [-3.14 to 0.09]

30. Secondary Outcome: Change From Baseline in Untrimmed Total Lung Volume With and Without Adjustment for Pre-BD FEV1
Description: as for outcome 25
Time Frame: Baseline and Week 13
Population: as for outcome 29
Measure: Mean (95% Confidence Interval); unit: Litre
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
Litre
  Untrimmed total lung volume at TLC: No adjustment for pre-BD FEV1 | 0.11 [-0.62 to 0.84]
  Untrimmed total lung volume at TLC: Adjusted for pre-BD FEV1 | 0.13 [-0.61 to 0.88]
  Untrimmed total lung volume at FRC: No adjustment for pre-BD FEV1: number analyzed (Participants) | 34
  Untrimmed total lung volume at FRC: No adjustment for pre-BD FEV1 | 0.52 [-0.16 to 1.21]
  Untrimmed total lung volume at FRC: Adjusted for pre-BD FEV1: number analyzed (Participants) | 34
  Untrimmed total lung volume at FRC: Adjusted for pre-BD FEV1 | 0.37 [-0.25 to 0.99]

31. Secondary Outcome: Change From Baseline in Untrimmed Total Mucus Volume Measured at TLC With and Without Adjustment for Pre-BD FVC
Description: The relationship between changes from baseline (week 0) in airway dynamics and conventional lung function measurements at Week 13, after accounting for baseline measurements of conventional lung function was assessed with and without adjustment for conventional lung function measures (pre-BD FVC).
Time Frame: Baseline and Week 13
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
mL
  No adjustment for pre-BD FVC | 0.05 [0.00 to 0.11]
  Adjusted for pre-BD FVC | 0.05 [-0.01 to 0.11]

32. Secondary Outcome: Change From Baseline in Untrimmed Total Mucus Plugs Score at TLC With and Without Adjustment for Pre-BD FVC
Description: Relationship between changes from baseline (week 0) in airway dynamics and conventional lung function measurements at Week 13, after accounting for baseline measurements of conventional lung function was assessed with and without adjustment for conventional lung function measures (pre-BD FVC). Mucus plugs was scored with a scoring system similar to that by Dunican et al. with SARP based on bronchopulmonary segmental anatomy. Mucus score was calculated by counting number of bronchopulmonary segments which contained 1 or more mucus plug, up to a maximum score of 18 corresponding to the 18 bronchopulmonary segments present in most people. In this system, a mucus plug is defined as a complete occlusion of airway visible at TLC. Each bronchopulmonary segment is given a score of 1 (mucus plug present) or 0 (mucus plug absent). The segment scores of each lobe are summed to generate a total mucus score for both lungs, yielding a mucus score ranging from 0-18. Higher scores = worse outcome.
Time Frame: Baseline and Week 13
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
Scores on a scale
  No adjustment for pre-BD FVC | 4.38 [-2.87 to 11.63]
  Adjusted for pre-BD FVC | 4.65 [-3.00 to 12.30]

33. Secondary Outcome: Change From Baseline in Untrimmed Total Air Trapping at FRC With and Without Adjustment for Pre-BD FVC
Description: as for outcome 31
Time Frame: Baseline and Week 13
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percentage of air trapping
Arm/Group | Benralizumab
Number analyzed (Participants) | 34
Percentage of air trapping
  No adjustment for pre-BD FVC | 3.18 [-3.65 to 10.01]
  Adjusted for pre-BD FVC | 4.36 [-2.06 to 10.79]

34. Secondary Outcome: Change From Baseline in Trimmed Distal Airway Wall Volume at TLC With and Without Adjustment for Pre-BD FVC
Description: as for outcome 31
Time Frame: Baseline and Week 13
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
mL
  No adjustment for pre-BD FVC | 5.29 [-1.39 to 11.97]
  Adjusted for pre-BD FVC | 6.08 [-0.60 to 12.76]

35. Secondary Outcome: Change From Baseline in Untrimmed Distal Airway Volume With and Without Adjustment for Pre-BD FVC
Description: as for outcome 31
Time Frame: Baseline and Week 13
Population: as for outcome 29
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
mL
  Untrimmed distal airway volume at TLC: No adjustment for pre-BD FVC | 2.20 [-1.09 to 5.49]
  Untrimmed distal airway volume at TLC: Adjusted for pre-BD FVC | 1.22 [-2.30 to 4.73]
  Untrimmed distal airway volume at FRC: No adjustment for pre-BD FVC: number analyzed (Participants) | 34
  Untrimmed distal airway volume at FRC: No adjustment for pre-BD FVC | -1.28 [-2.82 to 0.27]
  Untrimmed distal airway volume at FRC: Adjusted for pre-BD FVC: number analyzed (Participants) | 34
  Untrimmed distal airway volume at FRC: Adjusted for pre-BD FVC | -1.28 [-2.93 to 0.37]

36. Secondary Outcome: Change From Baseline in Untrimmed Total Lung Volume With and Without Adjustment for Pre-BD FVC
Description: as for outcome 31
Time Frame: Baseline and Week 13
Population: as for outcome 29
Measure: Mean (95% Confidence Interval); unit: Litre
Arm/Group | Benralizumab
Number analyzed (Participants) | 39
Litre
  Untrimmed total lung volume at TLC: No adjustment for pre-BD FVC | 0.11 [-0.62 to 0.84]
  Untrimmed total lung volume at TLC: Adjusted for pre-BD FVC | 0.11 [-0.63 to 0.85]
  Untrimmed total lung volume at FRC: No adjustment for pre-BD FVC: number analyzed (Participants) | 34
  Untrimmed total lung volume at FRC: No adjustment for pre-BD FVC | 0.52 [-0.16 to 1.21]
  Untrimmed total lung volume at FRC: Adjusted for pre-BD FVC: number analyzed (Participants) | 34
  Untrimmed total lung volume at FRC: Adjusted for pre-BD FVC | 0.40 [-0.22 to 1.02]

37. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The safety and tolerability of benralizumab was assessed.
Time Frame: From screening (Day -21) to follow-up (up to 1.9 years)
Population: The safety analysis set consisted of all participants who had received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab
Number analyzed (Participants) | 45
Participants
  Any AE | 17
  Any serious adverse event (SAE) | 2
  Any SAE with outcome death | 0
  Any AE leading to discontinuation of study intervention | 1
  Any possibly related AE | 3

ADVERSE EVENTS:
Time Frame: From screening (Day -21) to follow-up (up to 1.9 years)
Description: The Safety analysis set consisted of all participants who had received at least one dose of investigational product.
Arm/Group | Benralizumab
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 2/45
Other Adverse Events (participants affected / at risk) | 3/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab (N=45)
Respiratory tract infection (Infections and infestations) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab (N=45)
Gastroenteritis (Infections and infestations) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB.

DOCUMENTS (2):
  • Study Protocol (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT05552508/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT05552508/SAP_001.pdf